CLINICAL TRIAL: NCT05910372
Title: Development of Complementary Tools for the Differential Diagnosis of Fibromyalgia Based on Cognitive Task Performance
Brief Title: Tools for the Differential Diagnosis of Fibromyalgia Based on Cognitive Tasks
Status: Completed | Type: Observational
Sponsor: National Council of Scientific and Technical Research, Argentina (Other Government)
Collaborators: Center for Nuclear and Molecular Medicine Entre Ríos (Unknown)
Responsible Party: Principal Investigator, José Biurrun Manresa, PhD in Biomedical Science and Engineering, Advanced Bionics
Other Study IDs: IS003981
Record Dates: First submitted 2023-05-25; First posted 2023-06-18 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-10

CONDITIONS: Fibromyalgia
Keywords: Contralateral Delay Activity; Electroencephalography; Cognitive task; Biomarker
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Fibromyalgia Patients: Patients with primary fibromyalgia diagnosis. May include other chronic pain comorbidities, but the pain associated with those diseases should be less severe than the pain caused by fibromyalgia.
  Interventions: Other: Color Comparison Task; Other: N-back Task
- Healthy Controls: Volunteers with no clinical history of chronic pain, musculoskeletal or articular disorders.
  Interventions: Other: Color Comparison Task; Other: N-back Task

INTERVENTIONS:
Other: Color Comparison Task — Participants are presented with a series of colored squares and are instructed to compare the colors of two sequentially presented stimuli.
Other: N-back Task — Participants are presented with a sequence of letters and they must indicate whether the current stimulus matches the one presented 2 steps back in the sequence.

SUMMARY:
The goal of this observational study is to test for behavioural and neurophysiological biomarkers in fibromyalgia patients. The main questions it aims to answer are:

* Is there a measurable decline in working memory?
* Could these measures help in fibromyalgia differential diagnosis?

Participants will:

* perform Color Comparison tasks
* perform n-back tasks

DETAILED DESCRIPTION:
Fibromyalgia is a disease characterized by the presence of generalized musculoskeletal pain, accompanied by non-specific symptoms such as depression, sleep disturbances, anxiety, cognitive disabilities, among others. While widespread musculoskeletal pain is the predominant symptom in patients with fibromyalgia, cognitive impairments have also been widely reported, including decreased ability to concentrate, decreased short-term memory, and inability to multitask, which differentiate fibromyalgia patients from those with other chronic pain syndromes. Specifically, quantitative evidence has been found of impairment in executive functions in this group of patients, particularly in the domains of inhibitory control and working memory.

In the present study, participants (both healthy individuals and those diagnosed with fibromyalgia) will perform two cognitive tasks designed to assess the capacity and retrieval of information from working memory. The first task is the Color Comparison task, in which colored squares will appear on a computer screen for a short period of time. After a blank delay, a new set of squares will appear, and a decision has to be made about whether or not the squares are the same as the ones shown first. The task will be divided into 10 blocks of 30 trials each, with 10 trials comparing 2 colored squares, 10 trials comparing 4 colored squares, and 10 trials comparing 6 colored squares. A resting period will be given between each block. The behavioral results of this task will include reaction times and hit rates. At the same time, electroencephalographic data will be recorded to evaluate the Contralateral Delay Activity (CDA). The amplitude of this waveform is linked to the number of items allocated in working memory.

The second task that will be carried out by the participants is the n-back task. A sequence of letters will be presented, and participants will be asked to indicate whether the current stimulus matches the one presented two stimuli earlier. Sixty-two stimuli will be presented per block, and 5 blocks will be carried out. The results will be analyzed in terms of behavioral analysis and Event-Related Potentials (ERPs) analysis.

ELIGIBILITY:
Inclusion Criteria:

Fibromyalgia patients:

* Primary diagnosis of fibromyalgia according to the criteria used by the healthcare professional in charge of the patient.
* Other comorbidities are accepted as long as the pain caused by them is less severe than the pain caused by fibromyalgia.
* Willingness and ability to fully understand the content and scope of the experiment and to comply with the experiment instructions.
* Normal or corrected-to-normal vision.

Healthy controls:

* No history of neurological diseases, chronic pain or musculoskeletal disorders.
* Willingness and ability to fully understand the content and scope of the experiment and to comply with the experiment instructions.
* Normal or corrected-to-normal vision.

Exclusion Criteria:

Fibromyalgia patients:

* Pregnancy
* History of addictive behavior, defined as alcohol, cannabis, opioids or other drugs abuse.
* Presence of fever, tuberculosis, malignant tumors, infectious processes, acute inflammatory processes.
* Lack of cooperation

Healthy controls:

* Pregnancy
* History of chronic pain or musculoskeletal or articular disorders
* History of addictive behavior, defined as alcohol, cannabis, opioids or other drugs abuse.
* Presence of fever, tuberculosis, malignant tumors, infectious processes, acute inflammatory processes.
* Lack of cooperation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cohorts of patients and healthy controls wil be selected from the city of Paraná and surrounding areas. Through the ONG "Fibromialgia Entre Ríos Asociación Civil", the patients will be reached out and asked wether or not they are willing to participate. Additionally, flyer will be hung in major health facilities in the city and made public on social media. The cohort of healthy volunteers will be recruited after the patients for age, genre and socieconomic matching
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Percentage of correct answers in the Color Comparison task | Immediately after the intervention
  Percentage of correct answers over total number of trial in the Color Comparison Task

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire-Revised version (FIQR) | 10 minutes before the intervention
  Instrument for the assessment and evaluation of fibromyalgia patient's status
Symptoms Impact Questionnaire (SIQ) | 10 minutes before the intervention
  Instrument to assess healthy control's status regarding relevant clinical symptoms experienced in the last week.
Hospital Anxiety and Depression Scale (HADS) | 10 minutes before the intervention
  Widely used instrument to evaluate anxiety and depression
Brief Pain Inventory-Short Form (BPI-SF) | 10 minutes before the intervention
  It is an instrument to assess the severity of pain and its impact on functioning.
Power in EEG bands | Immediately after the intervention
  Analysis of EEG spectrum bands
Event-related potentials amplitude | Immediately after the intervention
  Amplitude, in microvolts, of event-related brain potentials
Event-related potentials latency | Immediately after the intervention
  Latency, in milliseconds, of event-related brain potentials

CONTACTS AND LOCATIONS:
Overall Officials: José A Biurrun Manresa, PhD, Principal Investigator — National Council of Scientific and Technical Research, Argentina (CONICET)
Locations (1):
- Center for Nuclear and Molecular Medicine Entre Ríos (CEMENER), Oro Verde, Entre Ríos Province, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be made available on the 'Open Science Framework' after undergoing the process of anonymization to remove any participant-identifying information. The data will consist of the raw EEG signals and raw behavioral responses to cognitive tasks. Additionally, the statistical analysis and Jupyter notebooks used to process the data will also be shared
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The participant's data and the processing pipeline will be available after the data collection is finished. The supporting information (including the study protocol, the statistical analysis plan and the informed consent) will be uploaded as soon as possible.
Access Criteria: The data will be publicly available.

REFERENCES:
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- [Background] Kravitz HM, Katz RS. Fibrofog and fibromyalgia: a narrative review and implications for clinical practice. Rheumatol Int. 2015 Jul;35(7):1115-25. doi: 10.1007/s00296-014-3208-7. Epub 2015 Jan 13. PMID 25583051
- [Background] Bell T, Trost Z, Buelow MT, Clay O, Younger J, Moore D, Crowe M. Meta-analysis of cognitive performance in fibromyalgia. J Clin Exp Neuropsychol. 2018 Sep;40(7):698-714. doi: 10.1080/13803395.2017.1422699. Epub 2018 Feb 1. PMID 29388512
- [Background] Adam KCS, Robison MK, Vogel EK. Contralateral Delay Activity Tracks Fluctuations in Working Memory Performance. J Cogn Neurosci. 2018 Sep;30(9):1229-1240. doi: 10.1162/jocn_a_01233. Epub 2018 Jan 8. PMID 29308988
- [Background] Shalchy MA, Pergher V, Pahor A, Van Hulle MM, Seitz AR. N-Back Related ERPs Depend on Stimulus Type, Task Structure, Pre-processing, and Lab Factors. Front Hum Neurosci. 2020 Oct 28;14:549966. doi: 10.3389/fnhum.2020.549966. eCollection 2020. PMID 33240059